CLINICAL TRIAL: NCT03861871
Title: Fenfluramine in CKDL5 Deficiency Disorder (CDD)
Brief Title: Fenfluramine in CDKL5 Deficiency Disorder (CDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-01530
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: CDD
Keywords: CKDL5 Deficiency Disorder
MeSH Terms: interventions — Fenfluramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fenfluramine Hydrochloride (Experimental): Study medication will be administered as equal doses twice a day in the morning and in the evening approximately 12 hours apart.
  Patients will first be titrated over 14 days to a dose of ZX008 0.8 mg/kg/day (maximum dose 30 mg/d).
  After completion of the Titration Period, patients will continue to receive the ZX008 0.8 mg/kg/day dose and be treated for an additional 12 weeks (Maintenance Period). Study medication will continue to be administered twice a day in the morning and in the evening, approximately 12 hours apart.
  After completion of the Maintenance Period, patients will enter the Taper Period, where they will decrease from 0.8 mg/kg twice a day to a dose of 0.4 mg/kg twice a day (maximum 30 mg/day). After 4 days at this dose level, patients will decrease their dose to 0.2 mg/kg/day. On day 9 of the Taper Period, all participants will stop taking study medication.
  Interventions: Drug: Fenfluramine Hydrochloride

INTERVENTIONS:
Drug: Fenfluramine Hydrochloride — Oral aqueous solution of fenfluramine hydrochloride buffered to pH 5 and provided in concentrations of 2.5 mg/mL. Manufactured by Andersonbrecon, Inc. on behalf of Zogenix International Limited.
  Other Names: ZX008

SUMMARY:
This study will be enrolling 10 patients, ages 2-18 years old, with a confirmed genetic/clinical diagnosis of CDKL5 Deficiency Disorder (CDD) in an open label trial of fenfluramine for seizure control. Patients will be titrated over 14 days to a dose of ZX008 0.8 mg/kg/day (maximum dose 30 mg/d).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical/genetic diagnosis of CDKL5 Deficiency Disorder CDD
* Ages 2-18 years old. Subject is male or non-pregnant, non-lactating female. Female subjects of childbearing potential must not be pregnant or breast-feeding. Female subjects of childbearing potential must have a negative urine pregnancy test. Subjects of childbearing or child-fathering potential must be willing to use medically acceptable forms of birth control, which includes abstinence, while being treated on this study and for 30 days after the last dose of study drug.
* Subject has been informed of the nature of the study and informed consent has been obtained from the legally responsible parent/guardian.
* Subject has provided assent in accordance with Investigational Review Board/Independent Ethics Committee (IRB/IEC) requirements, if capable.
* Subject's caregiver is willing and able to be compliant with diary completion, visit schedule and study drug accountability.
* Subjects must be receiving a therapeutically relevant and stable dose of anti-seizure medications, dietary therapies for epilepsy or vagus nerve stimulation settings for at least 4 weeks prior to screening and are expected to remain stable throughout the study.
* ≥4 convulsive seizures (tonic-clonic, tonic, atonic, clonic, focal motor) per 4-week period; each convulsive seizure must last ≥3 seconds.

Exclusion Criteria:

* Subject has a known hypersensitivity to fenfluramine or any of the excipients in the study medication.
* Subject has current or past history of cardiovascular or cerebrovascular disease, myocardial infarction or stroke.
* Subject has current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction or stroke, or clinically significant structural cardiac abnormality, including but not limited to mitral valve prolapse, atrial or ventricular septal defects, patent ductus arteriosis, and patent foramen ovale with reversal of shunt. (note: Patent foramen ovale or a bicuspid valve are is not considered exclusionary, but may be associated with the following diseases, which are exclusionary: coarctation of the aorta, Turner syndrome, supravalvular aortic stenosis, subvalvular aortic stenosis, patent ductus arteriosus, Sinus of Valsalva aneurysm, ventricular septal defect, Shone's complex, ascending aortic aneurysm, Loeys-Dietz syndrome, ACTA2 mutation familial thoracic aortic aneurysm syndrome, and MAT2A mutation familial thoracic aortic aneurysm syndrome).
* Subject has current or recent history of Anorexia Nervosa, bulimia, or depression within the prior year that required medical treatment or psychological treatment for a duration greater than 1 month.
* Subjects who are currently on CBD/THC or any MMJ or those who have tested positive urine tetrahydrocannabinol (THC) Panel or whole blood cannabidiol (CBD).
* Subject has participated in another clinical trial within the past 30 days (calculated from that study's last scheduled visit).
* Subject is at imminent risk of self-harm or harm to others, in the investigator's opinion, based on clinical interview.
* Subject has a current or past history of glaucoma.
* Subject is receiving concomitant therapy with: centrally-acting anorectic agents; monoamine-oxidase inhibitors; any centrally-acting compound with clinically appreciable amount of serotonin agonist or antagonist properties, including serotonin reuptake inhibition; atomoxetine, or other centrally-acting noradrenergic agonist; or cyproheptadine. (see appendix 1)
* Subject has moderate or severe hepatic impairment. Asymptomatic subjects with mild hepatic impairment (elevated liver enzymes <3x upper limited of normal [ULN] and/or elevated bilirubin <2x ULN) may be entered into the study after review and approval by the Medical Monitor in conjunction with the sponsor, in consideration of comorbidities and concomitant medications.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orrin Devinsky, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York Langone Health Comprehensive Epilespy Center, New York, New York, United States

REFERENCES:
- [Derived] Devinsky O, King L, Schwartz D, Conway E, Price D. Effect of fenfluramine on convulsive seizures in CDKL5 deficiency disorder. Epilepsia. 2021 Jul;62(7):e98-e102. doi: 10.1111/epi.16923. Epub 2021 May 12. PMID 33979451

RESULTS

PARTICIPANT FLOW:
Groups:
- Fenfluramine Hydrochloride: Study medication will be administered as equal doses twice a day in the morning and in the evening approximately 12 hours apart.
  Patients will first be titrated over 14 days to a dose of ZX008 0.8 mg/kg/day (maximum dose 30 mg/d).
  After completion of the Titration Period, patients will continue to receive the ZX008 0.8 mg/kg/day dose and be treated for an additional 12 weeks (Maintenance Period). Study medication will continue to be administered twice a day in the morning and in the evening, approximately 12 hours apart.
  After completion of the Maintenance Period, patients will enter the Taper Period, where they will decrease from 0.8 mg/kg twice a day to a dose of 0.4 mg/kg twice a day (maximum 30 mg/day). After 4 days at this dose level, patients will decrease their dose to 0.2 mg/kg/day. On day 9 of the Taper Period, all participants will stop taking study medication.
  Fenfluramine Hydrochloride: Oral aqueous solution of fenfluramine hydrochloride buffered to pH 5 and provided in concentrations of 2.5 mg/mL. Manufactured by Andersonbrecon, Inc. on behalf of Zogenix International Limited.
Period: Overall Study
Arm/Group | Fenfluramine Hydrochloride
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fenfluramine Hydrochloride
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Median Monthly Convulsive Seizure Frequency
Description: Change between baseline and Week 14 in the median number of monthly convulsive seizures.
Time Frame: Baseline, Week 14
Measure: Median (Standard Deviation); unit: Number of monthly seizures
Arm/Group | Fenfluramine Hydrochloride
Number analyzed (Participants) | 7
Number of monthly seizures | 88.429 (122.44)

2. Secondary Outcome: Change in Caregiver Global Impression of Change (CGIC) Score
Description: The CGIC is a 1-item, parent/caregiver-completed assessment used determine how much their child/care-recipient has improved with treatment. The instrument asks parents/caregivers to rate their child's/care-recipient's improvement as: 1) very much improved; 2) much improved; 3) minimally improved; 4) unchanged; 5) a little worse; 6) much worse; 7) very much worse; the total score correspondingly ranges from 1-7.
Time Frame: Baseline, Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fenfluramine Hydrochloride
Number analyzed (Participants) | 7
score on a scale | -2.429 (1.988)

3. Secondary Outcome: Change in Investigator Global Impression of Change (IGIC) Score
Description: The IGIC is a 1-item, investigator-completed assessment used determine how much a patient has improved with treatment. The instrument asks the investigator to rate patients' improvement as: 1) very much improved; 2) much improved; 3) minimally improved; 4) unchanged; 5) a little worse; 6) much worse; 7) very much worse; the total score correspondingly ranges from 1-7.
Time Frame: Baseline, Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fenfluramine Hydrochloride
Number analyzed (Participants) | 7
score on a scale | 1.571 (0.787)

4. Secondary Outcome: Change in Quality of Life in Childhood Epilepsy (QOLCE) Score
Description: Parent/caregiver-completed assessment assessing how epilepsy affects day-to-day functioning of their child/care-recipient in various life areas. Each item is ranked on a 5-point Likert scale from 1 (response correlated with the lowest possible quality of life) to 5 (response correlated with the highest possible quality of life). Item scores are then transformed to a 0-100 scale as follows: 1 = 0, 2 = 25, 3 = 50, 4=75, and 5=100. The total score is the average of all item scores and ranges from 0-100. Higher scores indicate greater quality of life; an increase in scores indicates quality of life increased during the observational period.
Time Frame: Baseline, Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fenfluramine Hydrochloride
Number analyzed (Participants) | 7
score on a scale | -0.429 (1.512)

5. Secondary Outcome: Change in Pediatric Quality Of Life (PEDS-QL) Epilepsy Module Raw Score
Description: The PedsQL Epilepsy Module is a 29-item measure with five scales: Impact, Cognitive, Sleep, Executive Function, and Mood/Behavior. The Impact scale (nine items) assesses how epilepsy interferes with daily activities, interacting with peers, independence, and increased disease burden due to treatment. The Cognitive Scale (six items) assesses memory, ability to learn new materials, school-related difficulties, and reading difficulties. The Sleep Scale (three items) assesses fatigue and sleep difficulties. The Executive Function Scale (six items) assesses organization, task initiation, impulsivity, and inattention. The Mood/Behavior Scale (five items) assesses feelings of anger, sadness, worries, and frustration tolerance. Scores range from 0-100 for each subscale, with higher scores representing better quality of life. The raw score is the sum of each subscale score and ranges from 0-500.
Time Frame: Baseline, Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fenfluramine Hydrochloride
Number analyzed (Participants) | 7
score on a scale | -103.571 (424.124)

ADVERSE EVENTS:
Time Frame: 14 Weeks
Description: Monitored via safety phone calls and at all visits.
Arm/Group | Fenfluramine Hydrochloride
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fenfluramine Hydrochloride (N=7)
Clostridium dificile infection (Infections and infestations) | 1
Respiratory infection (Infections and infestations) | 1
Aspiration pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fenfluramine Hydrochloride (N=7)
Diarrhea (Gastrointestinal disorders) | 2
Lethargy (General disorders) | 6
Crying episode (General disorders) | 2
Screaming episode (General disorders) | 1
Low appetite (General disorders) | 6
Upper respiratory infection (Infections and infestations) | 3
Common cold (Infections and infestations) | 3
Teething (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomitting (Gastrointestinal disorders) | 1
Weight Loss (General disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Pneumonia (Infections and infestations) | 1
Low grade fever (Infections and infestations) | 1
Bite on finger (General disorders) | 1
Intestinal gas (Gastrointestinal disorders) | 1
Grinding teeth (General disorders) | 1
Rash on face (General disorders) | 1
Hair loss (General disorders) | 1
Regurgitation after meals (Gastrointestinal disorders) | 1
Loose bowel (Gastrointestinal disorders) | 1
Low tone (General disorders) | 1
Loose stool (Gastrointestinal disorders) | 1
Mucus plug in throat (Infections and infestations) | 1
Irritability (General disorders) | 1
SARS-CoV2 infection (Infections and infestations) | 1
Sialorrhea (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT03861871/Prot_SAP_000.pdf